CLINICAL TRIAL: NCT03408522
Title: Clinical Characteristics and Functional Outcomes of Postoperative Myocardial Injury: A Prospective Cohort Study - Troponin Elevation After Major Noncardiac Surgery 2
Brief Title: Troponin Elevation After Major Noncardiac Surgery 2
Acronym: TEAMS2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Wilton A van Klei, Prof. dr., UMC Utrecht
Other Study IDs: TEAMS2
Record Dates: First submitted 2018-01-15; First posted 2018-01-24 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Perioperative Myocardial Infarction; Disability; Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Major adverse cardiac events (MACE) are a leading cause of mortality in patients undergoing noncardiac surgery. Patients with perioperative myocardial injury (PMI), defined as either myocardial infarction and lower elevations in cardiac troponin, are also at substantially increased risk of additional cardiac and noncardiac complications. Accordingly, it is plausible to assume that PMI negatively affects quality of life in terms of disability. The aim of this study is to investigate and compare the independent prognostic effects of the different PMI phenotypes (myocardial infarction and non-infarct troponin elevations) and noncardiac complications on disability in patients undergoing elective noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years old;
* Major noncardiac surgery defined as all noncardiac surgical procedures requiring an expected hospital stay of at least 24 hours;
* Elective surgery, defined as surgery that that has been preceded by a preoperative consultation at the anesthesia preoperative screening outpatient clinic.

Exclusion Criteria:

* Patients unable to fully comply to study needs (e.g. legally incapable patients or patients unable to communicate in Dutch or English).
* Patients with an American Society of Anesthesiologists (ASA) Physical status 5

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 years or older, undergoing major elective non-cardiac surgery under general or spinal anesthesia with an expected hospital admittance of at least 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Disability | 6 months after surgery
  Disability is expressed by the World Health Organization Disability Assessment Score 2.0 (WHODAS 2.0), which is based on difficulties experienced by the respondent in different functional domains including, cognition, mobility, self-care, getting along, life activities and participation during the previous 30 days. Disability is defined as a decrement in each functioning domain corresponding to score between 0% and 100%, in which no disability stands for a score of 0% and full disability represents a score of 100%, including death.

SECONDARY OUTCOMES:
Disability free survival | 6 months after surgery
  Disability free survival is defined as being alive with a WHODAS 2.0 score ≤ 25% and no increase of the pre-operative score ≥ 25% at 6 months after surgery.
Major adverse cardiovascular event (MACE) | 1 week after surgery
  MACE is defined as a composite outcome consisting of cardiovascular death, non-fatal myocardial infarction, non-fatal cardiac arrest, non-fatal ventricular fibrillation, ventricular arrhythmia with hemodynamic compromise, atrial fibrillation requiring cardioversion, pulmonary embolism, stroke
Noncardiac major adverse postoperative events (MAPE) | 1 week after surgery
  Noncardiac MAPE is a composite outcome consisting of respiratory failure (including pneumonia and hypoxia or hypercapnia leading to ICU admission for respiratory support), sepsis, renal failure, unplanned ICU admission, unplanned medium care admission, reoperation
Length of hospital stay | 1 week after surgery
  the number of days from the end of surgery until day of discharge
All-cause mortality | 1 week after surgery
Major adverse cardiovascular event (MACE) | 6 months after surgery
All-cause mortality | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wilton A van Klei, MD PhD, Principal Investigator — prof. dr.; W. Scott Beattie, MD PhD FRCPC, Principal Investigator — prof. dr.
Locations (3):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03408522/Prot_SAP_000.pdf